CLINICAL TRIAL: NCT00005996
Title: A Phase I Study of SU5416 in Combination With Gemcitabine/Cisplatin in Patients With Advanced Solid Tumors
Brief Title: SU5416 Combined With Gemcitabine and Cisplatin in Treating Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068000; UCLA-0002046; SUGEN-ND019901/SE5416.102; NCI-G00-1805
Record Dates: First submitted 2000-07-05; First posted 2004-07-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Gemcitabine; Semaxinib

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: semaxanib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. SU5416 may stop the growth of solid tumors by stopping blood flow to the tumor. Combining more than once chemotherapy drug with SU5416 may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of SU5416 combined with gemcitabine and cisplatin in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicities and pharmacokinetics of SU5416 when combined with gemcitabine and cisplatin in patients with advanced solid tumors. II. Determine the antitumor activity of this combination treatment regimen in this patient population.

OUTLINE: This is an open label, dose escalation study of SU5416. Patients receive gemcitabine IV over 30 minutes followed by cisplatin IV over 1 hour on day 1; SU5416 IV over 70 minutes on day 4; gemcitabine IV over 30 minutes followed by SU5416 IV over 70 minutes on day 8, and SU5416 on days 11, 15, and 18. Treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Following 6 courses of therapy, patients with stable and responsive disease may receive SU5416 alone on days 1, 4, 8, 11, 15, and 18 every 3 weeks for a maximum of 1 year. Cohorts of 3-6 patients receive escalating doses of SU5416 until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which at least one third of the patients experience dose limiting toxicity. Patients are followed at 1 month, and then every 3 months.

PROJECTED ACCRUAL: A total of 16-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced solid tumor that may respond to gemcitabine and cisplatin therapy (e.g., esophagus, head and neck, breast, ovary, bladder, or non-small cell lung cancer) No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8.8 g/dL Hepatic: Bilirubin less than 2.05 mg/dL Renal: Creatinine no greater than 1.8 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: No prior myocardial infarction No severe or unstable angina No history of atherosclerotic coronary artery disease requiring coronary or peripheral artery bypass surgery or concurrent medication No history of arrhythmias, hypertension, or deep venous thrombosis No clinical evidence of severe peripheral vascular disease related to diabetes mellitus Pulmonary: No history of lung embolism Other: No known allergy to Cremophor or Cremophor based drug products No contraindications to systemic gemcitabine or cisplatin therapy No insulin dependent or noninsulin dependent diabetes mellitus with clinical evidence of diabetic ulcers No other active malignancies except basal cell skin cancer or carcinoma in situ of the cervix No other acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 weeks since prior epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF) No prior antiangiogenesis therapy No prior SU5416 No concurrent immunotherapy Chemotherapy: See Disease Characteristics No more than 1 prior systemic chemotherapy regimen allowed At least 4 weeks since prior systemic chemotherapy (6 weeks for mitomycin or nitrosourea) No prior high dose chemotherapy At least 6 months since prior gemcitabine and cisplatin and responsive No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: At least 4 weeks since prior surgery Other: No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Rosen, MD, Study Chair — Jonsson Comprehensive Cancer Center